CLINICAL TRIAL: NCT02024256
Title: Comparison Between Treatment With Gauze Soaked With Cold Magnesium Sulfate Solution Against Gauze Soaked With Cold Water for Treatment of Perineal Swelling Following Vaginal Delivery - A Double Blind Placebo Controlled Trial
Brief Title: Cold Magnesium Sulfate Solution for Perineal Swelling Following Vaginal Delivery
Acronym: MgSo4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MG33
Record Dates: First submitted 2013-12-25; First posted 2013-12-31 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Vaginal Delivery; Perineal Swelling; Perineal Pain
Keywords: Vaginal delivery; Perineal swelling; Perineal pain; MgSo4; Magnesium sulfate; Cold water
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium sulfate (Active Comparator): Pads soaked in cold magnesium sulfate solution
  Interventions: Other: Cold pads soaked in Magnesium sulfate solution
- Water (Sham Comparator): Pads soaked with cold water
  Interventions: Other: Cold pads soaked in water

INTERVENTIONS:
Other: Cold pads soaked in Magnesium sulfate solution
  Other Names: Epson salt, MgSo4
  Arms: Magnesium sulfate
Other: Cold pads soaked in water
  Arms: Water

SUMMARY:
The purpose of this study is to compare the impact of treatment with cooled magnesium sulfate and cold water-soaked pads on perineal pain and swelling following vaginal delivery.

Assessment of appropriateness for each patient to take part in the study will be performed approximately 2 hours following delivery. Those patients who consent to participate in the trial will be allocated to treatment groups in a double-blinded, randomized manner. Women in the study group will receive treatment with pads soaked in a cold aqueous solution of magnesium sulfate at 33% (w/v) concentration, while those in the control group will receive treatment with pads soaked in cold water.

Nurses will initiate treatment according to the group to which the patient was randomized. Said pads will be given the patients routinely 5 times a day at regular times.

A physician will assess the perineal swelling according to visual (photographed) scale in which severe, moderate, light and no swelling will be defined. Measurement of swelling in centimeters (maximal length and breadth); photography, by a medical photographer or the examining doctor, of the perineal area with a centimeter ruler, before, during and after treatment (photography is dependent on patient approval and is not a precondition to participation in the trial.); and additional examination, on the above basis, will be performed regarding hemorrhoids in the event that a patient has complained of such.

A nurse will assess the perineal pain and swelling on a scale ranging from 0 to 10 prior to the patient being given the pad and an hour following treatment. An additional assessment by the same method will be performed regarding hemorrhoid pain. Any analgesia administered will also be recorded.

Likewise, for follow-up purposes a blood test for serum magnesium concentration will be taken before and after treatment.

Period of follow-up will be 48-72 hours from childbirth.

ELIGIBILITY:
Inclusion Criteria:

* parturients following normal vaginal birth or vacuum-assisted vaginal delivery
* reporting of perineal pain equal to or greater than 3 on a 0-10 scale

Exclusion Criteria:

* parturients following cesarean section
* lack of consent to take part in the study
* parturients interested in early discharge (within 48 hours of childbirth)
* girls under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the level of perineal pain | 3 days
Reduction in perineal swelling | 3 days

SECONDARY OUTCOMES:
Reduction in hemorrhoids pain and swelling | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Nahum, MD, Principal Investigator — HaEmek medical center affiliated to Rappaport faculty of medicine, Technion, Haifa, Israel
Locations (2):
- Israel (2):
  - HeEmek medical center, Afula
  - HaEmek medical center, Afula

REFERENCES:
- [Derived] East CE, Dorward ED, Whale RE, Liu J. Local cooling for relieving pain from perineal trauma sustained during childbirth. Cochrane Database Syst Rev. 2020 Oct 9;10(10):CD006304. doi: 10.1002/14651858.CD006304.pub4. PMID 33034900